CLINICAL TRIAL: NCT05282589
Title: Effects Of Lumbopelvic Manipulation On Fatigue In Chronic Low Back Pain Patients
Brief Title: Lumbopelvic Manipulation Effects on Fatigue in Chronic Low Back Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rphah/RCRS/REC/01057
Record Dates: First submitted 2022-02-20; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Intervention Model Description: parallel assignment
Who Masked: Participant
Masking Description: single blinded means that the participants have no idea of what treatment they are receiving and to which group they belong.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumbopelvic manipulation and conventiontional therapy (Experimental): Group A an experimental group was given conventional therapy and lumbopelvic manipulation. conventional therapy include TENS and Hot pack for 20 minutes , hamstrings stretching, calf stretching,transversus abdominis strengthening and lumber multipedes muscle strengthening. while lumbopelvic manipulation include high velocity thrust given in posterior direction to ASIS.
  Interventions: Other: lumbopelvic manipulation and conventional therapy
- conventional therapy (Active Comparator): Group B, control group was given only conventional therapy which include TENS and Hot pack for 20 minutes , hamstrings stretching, calf stretching,transversus abdominis strengthening and lumber multipedes muscle strengthening . 1 set of 10 repetitions, 3 sessions per week with a total of 12 sessions.
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: lumbopelvic manipulation and conventional therapy — Lumbopelvic manipulation was given along with conventional physical therapy
  Transcutaneous Electrical Nerve Stimulation was applies for 15 minutes. 3 alternate days per week.
  Static stretching exercises for targeted muscles Erector spinae, hamstrings and calfs) - 4 repetations X 2 sets with 30 seconds hold and 1 minute of resting interval. On 03 alternate days per week.
  Strengthening exercises for traverses abdomminis and lumber multipedus muscles - 15 repetitions X 3 sets. On 03 alternate days per week.
  Total 12 session were given, each consisting of 45 minutes.
  Arms: Lumbopelvic manipulation and conventiontional therapy
Other: conventional therapy — Transcutaneous Electrical Nerve Stimulation was applies for 15 minutes. 3 alternate days per week.
  Static stretching exercises for targeted muscles Erector spinae, hamstrings and calfs) - 4 repetations X 2 sets with 30 seconds hold and 1 minute of resting interval. On 03 alternate days per week.
  Strengthening exercises for traverses abdomminis and lumber multipedus muscles - 15 repetitions X 3 sets. On 03 alternate days per week.
  Total 12 session were given, each consisting of 45 minutes.
  Arms: conventional therapy

SUMMARY:
The aim of the study is determine the effects of lumbopelvic manipulation on fatigue, pain and disability in chronic low back pain patients. In this randomised clinical trial, lumbopelvic manipulation group was compared with conventional therapy group. Tools used in the study are numeric pain rating scale ,oswestry low back pain index and rating of fatigue scale.

DETAILED DESCRIPTION:
Low back pain is an extremely common problem which causes morbidity in adults. It is more likely to occur in individuals around the age 20 to 60, this is partly due to the changes that occurs with aging. It can be acute (less than 12 weeks) or chronic (more than 12 weeks). There are many causes of low back pain one of the most common is the lumber disc herniation. Some of the most serious causes of low back pain include (infection, malignancy, vertebral fracture, cauda equina syndrome and inflammatory disorders such as axial spondyloarthritis). Mostly low backpain can be a result of injury such as muscle strain or sprains due to sudden movements or poor body mechanics while lifting heavy loads. Pain in low back can be the result of infection effecting the bony lumber spine, ligaments around the spine, the spinal cord, nerves and muscles of the spine, internal organs and skin around the spine.

Treatment for low back pain falls into three broad categories, multidisciplinary therapy is based on intensive exercises that improves physical function and has modest effects on pain physiotherapy treatment of low back pain includes laser, massage, multidisciplinary rehabilitation and spinal manipulation. Spinal manipulation is a high velocity thrust to a joint beyond its restricted range of movement. Spinal manipulation to lumber spine is a common intervention administered for patients with low back pain.

There is limited use of the technique in our society especially finding its effects on fatigue in chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

females patients having fatigue along with chronic low back pain low back pain for more than three months age 20-60

Exclusion Criteria:

* patients with conditions other than chronic low back pain having radiculopathy history of serious underlying pathology such as nerve root compromise, structural deformities, genetic spinal disorders and previous spinal surgery.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Fatigue assessment scale (FAS) | 4th week
  Among the ten questions of the FAS. Every point of has further five components in which 1 means "never" and 5 means "always". Its scoring is from 10-50 in which 10 showing lowest fatigue level and 50 means indicating highest fatigue level.
  If the overall score is less than 22 it denotes no fatigue while if the score is more than 22 it will show the presence of substantial fatigue.

SECONDARY OUTCOMES:
Numeric pain rating scale (NPRS) | 4th week
  Numeric pain rating scale is 11 point scale which consists of a straight or linear line running from left to right with a range from 0 -10 in which the digit 0 which lies on the left means no pain while the digit 10 lying on the right means the worst pain.
Oswestry low back pain questionnaire | 4th week
  The oswestry low back pain questionnaire is believed to be specially designed for back related disability in daily life activities in 10 queries with a substitutes for verbal response. Its ranking is from 0-100 in which 0 means there is no disability at time and 100 score means absolutely or entirely disabled.
Range of Motion | 4th week
  It was measured by bubble inclinometer. For taking the ranges of flexion and extension 12th thoracic and 1st sacral vertebrae were taken as the reference points. Two bubble inclinometers were used at the same time in standing position.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Affan Iqbal, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No